CLINICAL TRIAL: NCT04818294
Title: Prospective, Multi-center, Clinical Trial (Phase IV Study) to Monitor the Efficacy of Treatment by Applying a High Electrostatic Charge to Patients With Chronic Pain, in the Practice of Clinical or Out-patient Pain Treatment Facilities.
Brief Title: Clinical Trial to Monitor the Efficacy of the Elosan Treatment by Applying Electrostatic
Status: Completed | Type: Observational
Sponsor: Elosan AG (Industry)
Responsible Party: Sponsor
Other Study IDs: ELES_03
Record Dates: First submitted 2021-03-19; First posted 2021-03-26 (Actual); Last update posted 2023-01-26 (Actual); Status verified 2023-01

CONDITIONS: Chronic Pain
MeSH Terms: conditions — Chronic Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Pain treatment by electrostatic charge to the whole body — Study Type is Observational as participants in the study receive therapeutic interventions in the therapy cabin as part of routine medical care and a researcher studies the effect of the intervention.
  The study includes all persons who are already receiving therapy in the mentioned facilities, no external, specifically selected persons, but existing patients suffering from chronic pain who meet the specified conditions.
  The therapy aims to alleviate chronic pain by applying an electrostatic charge of 50'000 Volt to the whole body in the special, electrically insulated cabin. The treatment is done upon the instructions of a physician. It is done with the patient standing up in the treatment cabin. The person is charged and discharged several times over the course of 2x 4 minutes. The charge can be felt on the skin and it can be seen through bristling of the hairs on the body. This treatment is repeated once a week.

SUMMARY:
The Treatment Cabin 'Elosan cabin' is a closed, electrically insulated cabin for the short-term application of a high electrostatic voltage to the body of patients with chronic pain.

Patients assigned will have 8 sessions in the treatment cabin, with an interval of 6 days between sessions. The existing therapies and painkillers will be continued at the discretion of the doctor.

DETAILED DESCRIPTION:
Included in the study can be all persons suffering from chronic pain as it is often the case with rheumatic disease or traumata. The electric charge is created by a generator which can produce a high electrostatic field. The electrical voltage is delivered to the hands via a metal handle and is spread over the entire body surface. After the short treatment, the patient is completely discharged and earthed again.

Over 100 patients in eight pain centers are to be included into this trial in order to show a statistically significant reduction of pain.

ELIGIBILITY:
Inclusion Criteria:

* Informed Consent
* adults, age ≥ 18 years, male or female patients
* History of pain ≥ 3 months
* Suffering from chronic pain
* Intensity of pain rated ≥ 50 mm on VAS pain

Exclusion Criteria:

* Patients with an electrical or electronic implant.
* Women who are pregnant, breastfeeding or planning to become pregnant
* Patients who have already been treated with the cabin within the last 4 weeks.
* Patients who are currently participating in other studies or who have participated in other studies in the last 30 days
* Patients who have indicated their intention or who are suspected of intending to discontinue or discontinue therapy before the end of the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study will include pain patients who are already being treated in the practice of clinical or resident pain therapy facilities.
Sampling Method: Probability Sample
Enrollment: 192 (Actual)
Dates: Start 2021-03-16 (Actual); Primary Completion 2022-05-15 (Actual); Study Completion 2022-06-15 (Actual)

PRIMARY OUTCOMES:
Change of Pain Intensity is being assessed by Visual Analogue Scale (VAS) | 8-9 weeks
  Change of Pain Intensity is being assessed on a horizontal 100 mm VAS (Visual Analogue Scale) pain scale. The total range of this scale is 100 mm. Minimum score is 0 mm, Maximum score is 100 mm. The higher values represent a higher intensity of pain. The values at baseline will be compared to the values at Visit 8 and the mean of the differences will be compared between the 2 treatment arms.

SECONDARY OUTCOMES:
Composite outcome physical health (PCS) and mental health (MCS) to determine the quality of life assessed by the SF-12 Questionnaire | 8-9 weeks
  Patients fill out a 12 question survey at the first and the last visit, which is then scored by a researcher.
  The 12-Item Short Form Survey (SF-12) is designed as a general measure of health. It is a quality of Well-Being Score in comparison to US general population. Composite outcome physical health (PCS) and mental health (MCS) to determine the quality of life assessed by SF-12 Questionnaire compared to the United States average (avg=50)
  The change in quality of life (as reported by SF 12 questionnaires) from baseline to end of treatment (Day 28) will be compared between the treatment groups. The impact of the changes in summary scores (NBS: Norm-Based-Scoring) of physical health (PCS) and mental health (MCS) will be assessed by a General Linear Model (GLM) using the treatment as fixed factors and the baseline PCS and MCS as covariates, respectively.
Pain medication / therapy and any changes thereof shall be recorded during the study. | 8-9 weeks
  To determine the effects on standard treatment, medication and other, different therapies, a special questionnaire is collected per patient.
  This lists the dose of all medications and therapies as follows:
  * until the start of the study
  * at each of the 8 visits
  * at the end of the study
  Medication will vary from patient to patient. Therefore, the dose of comparable medications/therapies, mainly pain medications, will be assessed.
  The pain medication taken at baseline will be compared to the amount of pain medication taken at the end of treatment. Changes in pain medication will be qualified by the investigators as either being clinically relevant or not.

OTHER OUTCOMES:
Improving the quality of sleep | 8-9 weeks
  The quality of sleep is recorded on the questionnaire at each visit

CONTACTS AND LOCATIONS:
Overall Officials: Stephan Steinhauser, M.D., Principal Investigator — Stadtspital Triemli, 8063 Zürich
Locations (8):
- Switzerland (8):
  - Centro Ortho-Bio-Med, Roveredo, CH
  - Zentrum für Neurochirurgie Hirslanden Ostschweiz, Sankt Gallen, CH
  - Medizinisches Zentrum, Bad Ragaz
  - Spital Emmental, Schmerzzentrum, Burgdorf
  - Rheumapraxis Cham Zug, Cham
  - Praxis Dr. Kessler, Lucerne
  - Orthopädische Schmerztherapie Zürich, Zurich
  - Schulthess Klinik Zürich, Zurich

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Steinhauser S, Ganter MT, Stadelmann V, Hofer CK; ELES Study Group. Whole-Body Electrostatic Pain Treatment in Adults with Chronic Pain: A Prospective Multicentric Observational Clinical Trial. Pain Ther. 2024 Feb;13(1):69-85. doi: 10.1007/s40122-023-00560-8. Epub 2023 Nov 28. PMID 38015366